CLINICAL TRIAL: NCT02096146
Title: TMT Fusion Plate vs. Two Crossed Screws - A Randomized Controlled Trial
Brief Title: TMT Fusion Plate vs. Two Crossed Screws
Acronym: TMT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrolment
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMT Fusion Plate
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Clinical Indication for First Metatarsal Joint Arthrodesis
Keywords: Plate; Hallux valgus; Foot deformity; Screw; Tarsometatarsal angle; Cost effectiveness
MeSH Terms: conditions — Hallux Valgus; Foot Deformities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMT Fusion Plate (Other): Patients are treated with TMT Fusion Plate to encourage bony fusion of the 1st TMT joint.
  Interventions: Procedure: TMT Fusion plate
- Two crossed screws (Other): Patients are treated with two crossed screws.This procedure is a standard treatment for 1st TMT joint fusion .
  Interventions: Procedure: Two crossed screws

INTERVENTIONS:
Procedure: TMT Fusion plate — Patients are treated with TMT Fusion Plate a post-market device to encourage bony fusion of the 1st TMT joint.
  Arms: TMT Fusion Plate
Procedure: Two crossed screws — Patients are treated with two crossed screws.This procedure is a standard treatment for 1st TMT joint fusion.
  Arms: Two crossed screws

SUMMARY:
This study will compare TMT Fusion Plate versus two crossed screws for the fixation of first tarsometatarsal joint arthrodesis. Patients who meet eligibility criteria will be randomly assigned to one of these two treatment options.

DETAILED DESCRIPTION:
Tarsometatarsal joint arthrodesis is a common procedure which can be performed using various devices such as screws, plates or both. The Tarsometatarsal Fusion Plate from "DePuySynthes" is a new device designed to encourage bony fusion of the 1st TMT joint, and is expected to lead to earlier fusion compared to the current standard of care of using 2 crossed screws. This is expected, in turn, to result in an earlier reduction in pain and an earlier return to full activity. At this time there is insufficient data directly comparing outcome following surgery for patients treated with screws or plates, and a study protocol which produces a higher level of evidence is therefore necessary.

The main aim of this study is to compare patient-reported outcome following surgery for patients undergoing joint arthrodesis using the TMT Fusion plate versus screws only. It is expected that surgery will improve patient-reported outcome similarly for both treatment groups in the long-term, but that the improvement will occur earlier for the plate group. For this study patient-reported outcome will be assessed by the walking/standing and pain domain scores of the Manchester Oxford Foot Questionnaire (MOXFQ). An earlier improvement in any of these two domains would be considered to be valuable. The primary analysis will therefore compare the time to a minimal clinically relevant improvement for any of the two MOXFQ domains for patients treated with TMT fusion plate versus patients treated with only screws during the first 12 months following surgery.

An economic evaluation from a societal perspective will determine the incremental cost-effectiveness of the TMT fusion plate versus the 2 crossed screws technique for 1st TMT joint fusion. Therefore a randomized controlled trial will be conducted, where patient-reported outcomes as well as clinical outcome parameters will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 65 years
* At least one of the following:

  * 1st TMT arthritis
  * hallux valgus (intermetatarsal angle (IM) 1-2 angle > 15° on plain x-ray)
  * 1st ray hypermobility with or without flat foot
* Painful condition
* Ability to understand the content of the patient information / Informed Consent Form
* Willingness and ability to participate in the clinical investigation according to the Clinical Investigation Plan (CIP)
* Signed and dated IRB/EC-approved written informed consent

Exclusion Criteria:

* Active infection
* Previous surgery on the 1st ray of the same foot
* Previous non-union on the 1st ray of the same foot
* Clinical obvious arthritis in other joints of the lower extremities
* Purely seeking plastic surgery
* Peripheral vascular disease (e.g. advanced diabetes)
* Peripheral sensory neuropathy (e.g. advanced diabetes)
* Concurrent surgery of the contralateral foot
* Any previously medically unmanaged severe systemic disease
* Substance abuse that would preclude reliable assessment
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in the patient-reported MOXFQ | Up to 4 weeks pre-operative, Discharge (up to 1 week post-operative), 2 week FU, 6 week FU, 3 month FU, 6 month FU, 12 month FU
  Outcome measures for the study focus on fully validated patient related outcome measures for the foot (MOXFQ).

SECONDARY OUTCOMES:
Development of bone healing assessed based on x-rays | 6 and 12 weeks postoperative
Reconstruction of the joint position based on x-rays | Pre-operative up to 4 weeks vs. post-operative up to 2 weeks
Change in quality of life (EQ-5D) | Up to 4 weeks pre-operative, discharge (up to 1 week post-op), 2 weeks FU, 6 weeks FU, 3 months FU, 6 months FU, 12 months FU
  Outcome measure of general health
Weekly assessed weight bearing during weeks 6-12 | 3 months FU
Complications related to implant or surgery | Starts with surgery and is continued until the end of the study (12 months FU)
  For the duration of the study complications are continuously recorded and not restricted to the defined follow up visits.
Documentation of medication and treatment costs | Starts after surgery and is continued until the end of the study (12 months FU)
  A cost diary to collect treatment costs is distributed and collected at the next FU visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Winson, MB ChB, FRCS, Principal Investigator — Southmead Hospital
Locations (5):
- United States (3):
  - Mid Michigan Orthopedic Institute - East Lansing, East Lansing, Michigan
  - Summit Orthopedics, Woodbury, Minnesota
  - NY Downtown Orthopedic Associates, New York, New York
- Centro Médico Imbanaco Cali, Cali, Colombia
- Ian Winson, Bristol, United Kingdom